CLINICAL TRIAL: NCT03570320
Title: Does Altering Narcotic Prescription Methods Affect Opioid Distribution Following Select Upper Extremity Surgeries?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Yanik (Other)
Responsible Party: Sponsor-Investigator, John Yanik, Resident Physician, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201804820
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Opioid Use
Keywords: opioid; narcotic; postoperative; prescription; refill; upper extremity surgery

STUDY DESIGN:
Intervention Model Description: Control arm versus interventional arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The first treatment group will be our control arm. On discharge following their surgery, these patients will receive a single prescription for 225 Morphine Milligram Equivalents (MMEs). This corresponds to #30 pills of 5mg oxycodone/acetaminophen, #45 pills of 5mg hydrocodone/acetaminophen, or #30 pills of 7.5mg Morphine.
- Interventional Arm (Experimental): Patients who are randomized into the second group will also receive prescriptions for 225 MME's on discharge following their surgery, however their medications will be broken up equally into 3 separate scripts, each for 75 MME's. This corresponds to 3 scripts for #10 pills of 5mg oxycodone/acetaminophen, 3 scripts for #15 pills of 5mg hydrocodone/acetaminophen, or 3 scripts for #10 pills of 7.5mg Morphine. Each script will be post-dated to ensure that patients wait the appropriate amount of time between filling their scripts, and that they cannot fill multiple scripts on the same day or at the same time.
  Interventions: Other: Modification of opioid prescription method

INTERVENTIONS:
Other: Modification of opioid prescription method — Patients in the interventional arm of the study will receive post-op opioid medications in three small prescriptions as opposed to one large prescription. They may fill these prescriptions as needed.
  Arms: Interventional Arm

SUMMARY:
It has been well established that prescription opioid misuse and prescription opioid abuse is on the rise. In the late 1990's and early 2000's, there was a large push to make "pain" the fifth vital sign. At the same time, direct-to-consumer advertising and changes in national guidelines laid the groundwork for a decade that would ultimately see the amount of narcotic prescriptions in the United States more than double, and the number of prescription-opioid related deaths more than quadruple.

Recently, providers have started to question their own role in this epidemic. In the field of orthopedics in particular, considerable emphasis is now being placed on developing a better understanding of patients postoperative pain requirements, and amending practices to continue to meet those requirements while at the same time responsibly limiting the amount of narcotics that are prescribed. The goal of this project is to further this line of research by testing an opioid prescription model that is designed to easily reconcile clinical practices for prescribing pain medications with individual patient needs.

The investigators propose to evaluate a new method for prescribing opioid pain medications that consists of giving patients smaller amounts of narcotics with easier access to refills. It is hypothesized that in this system, patients will ultimately obtain fewer pills from the pharmacy, and will have fewer pills left over following their post-operative recovery. To test this hypothesis, a randomized controlled trial has been designed wherein patients will be given either one single prescription for opioid medications (control group, representing current practice) or multiple small prescriptions for opioid medications that they may fill on an as-needed basis (intervention group). The total amount of narcotics prescribed to both groups will be the same; only the number of prescriptions and the size of each prescription will be altered.

Unused narcotic medications are ripe for diversion and may potentially be playing a significant role in the opioid abuse crisis that we are experiencing in the United States. Developing strategies to minimize left over pills while maintaining adequate pain control is perhaps one of the most crucial first steps in addressing this important issue. The success of this model could have broad implications across the healthcare profession. From surgery to emergency medicine and even primary care, this model would be easy to implement and may provide an effective way for the medical community to start to combat the opioid epidemic.

DETAILED DESCRIPTION:
The investigators propose to evaluate a method for prescribing opioid pain medications in the acute post-operative period. This approach consists of giving patients smaller amounts of narcotics with easier access to refills. The investigators hypothesize that in this system, patients will ultimately obtain fewer pills from the pharmacy, and will have fewer pills left over following their post-operative recovery. To test this hypothesis, a randomized controlled trial has been designed. The investigators have chosen patients undergoing open reduction and internal fixation of distal radius fractures and patients undergoing first carpometacarpal joint arthroplasty as the study population. In the literature, the investigators experience, anecdotally, and as was demonstrated with a brief informal survey that was collected, these groups of patients have similar opioid needs postoperatively, and that need is relatively high when compared to other hand and upper extremity surgeries.

Intervention:

Patients will be consented on the day of surgery. Patients who consent in the preoperative area will be sequentially randomized to one of two treatment groups. The first treatment group will be the control arm. On discharge following their surgery, these patients will receive a single prescription for 225 Morphine Milligram Equivalents (MMEs). This corresponds to #30 pills of 5mg oxycodone/acetaminophen, #45 pills of 5mg hydrocodone/acetaminophen, or #30 pills of 7.5mg Morphine.

Patients who are randomized into the second group will also receive prescriptions for 225 MME's on discharge following their surgery, however their medications will be broken up equally into 3 separate scripts, each for 75 MME's. This corresponds to 3 scripts for #10 pills of 5mg oxycodone/acetaminophen, 3 scripts for #15 pills of 5mg hydrocodone/acetaminophen, or 3 scripts for #10 pills of 7.5mg Morphine. Each script will be post-dated to ensure that patients wait the appropriate amount of time between filling their scripts, and that they cannot fill multiple scripts on the same day or at the same time. Patient consent, randomization, surgery, and discharge with their scripts will all occur on the day of their operation.

Should a patient call in or come to clinic requesting more narcotic medication, the study policy will be that all patients are eligible to receive additional scripts in increments of 75 MME's regardless of their initial randomized group (an additional #10 pills of 5mg oxycodone/acetaminophen, #15 pills of 5mg Hydrocodone/acetaminophen, or #10 pills of 7.5mg Morphine). The number of additional scripts that patients may receive will be at the discretion of the surgeon who performed the procedure. Patients will have to make separate requests for each additional script - the investigators will not give multiple additional scripts at once. If the physician and patient feel that it is in the patient's best interest, they may transition from one narcotic to another at the time of a refill.

The investigators will assess the patients post-operative narcotic use including the number of pills distributed from the pharmacy to each group, number of pills consumed, and number of pills retained after the patient is no longer requiring them. The investigators will also assess patients general pain control, comfort level, and standard outcomes during the recovery period.

ELIGIBILITY:
Inclusion Criteria:

* Patients at the University of Iowa Hospitals and Clinics will be eligible for this study if they are over the age of 18 and are undergoing outpatient ORIF of isolated unilateral distal radius fractures or first CMC joint arthroplasty.

Exclusion Criteria:

* Patients will be excluded if they are undergoing surgery for an infection, receiving revision surgery, have multiple injuries that require narcotic use, have a history of chronic narcotic use, or cannot provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Number of pills dispensed from a pharmacy to patients | For each patient, this outcome will be assessed out to 8 weeks postoperatively or when the patient is no longer requiring pain medications.
  Investigators will track how many pills were dispensed from a pharmacy to patients in each group.

CONTACTS AND LOCATIONS:
Overall Officials: John M Yanik, MD, Principal Investigator — University of Iowa Hospitals and Clinics, Department of Orthopedics and Rehabilitation
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brat GA, Agniel D, Beam A, Yorkgitis B, Bicket M, Homer M, Fox KP, Knecht DB, McMahill-Walraven CN, Palmer N, Kohane I. Postsurgical prescriptions for opioid naive patients and association with overdose and misuse: retrospective cohort study. BMJ. 2018 Jan 17;360:j5790. doi: 10.1136/bmj.j5790. PMID 29343479
- [Background] Caudill-Slosberg MA, Schwartz LM, Woloshin S. Office visits and analgesic prescriptions for musculoskeletal pain in US: 1980 vs. 2000. Pain. 2004 Jun;109(3):514-519. doi: 10.1016/j.pain.2004.03.006. PMID 15157714
- [Background] Clark DJ, Schumacher MA. America's Opioid Epidemic: Supply and Demand Considerations. Anesth Analg. 2017 Nov;125(5):1667-1674. doi: 10.1213/ANE.0000000000002388. PMID 29049112
- [Background] Dwyer MK, Tumpowsky CM, Hiltz NL, Lee J, Healy WL, Bedair HS. Characterization of Post-Operative Opioid Use Following Total Joint Arthroplasty. J Arthroplasty. 2018 Mar;33(3):668-672. doi: 10.1016/j.arth.2017.10.011. Epub 2017 Oct 16. PMID 29128235
- [Background] Florence CS, Zhou C, Luo F, Xu L. The Economic Burden of Prescription Opioid Overdose, Abuse, and Dependence in the United States, 2013. Med Care. 2016 Oct;54(10):901-6. doi: 10.1097/MLR.0000000000000625. PMID 27623005
- [Background] Jones CM, Paulozzi LJ, Mack KA. Sources of prescription opioid pain relievers by frequency of past-year nonmedical use United States, 2008-2011. JAMA Intern Med. 2014 May;174(5):802-3. doi: 10.1001/jamainternmed.2013.12809. No abstract available. PMID 24589763
- [Background] Kim N, Matzon JL, Abboudi J, Jones C, Kirkpatrick W, Leinberry CF, Liss FE, Lutsky KF, Wang ML, Maltenfort M, Ilyas AM. A Prospective Evaluation of Opioid Utilization After Upper-Extremity Surgical Procedures: Identifying Consumption Patterns and Determining Prescribing Guidelines. J Bone Joint Surg Am. 2016 Oct 19;98(20):e89. doi: 10.2106/JBJS.15.00614. PMID 27869630
- [Background] Levin P. The Opioid Epidemic: Impact on Orthopaedic Surgery. J Am Acad Orthop Surg. 2015 Sep;23(9):e36-7. doi: 10.5435/JAAOS-D-15-00250. Epub 2015 Aug 13. No abstract available. PMID 26271757
- [Background] Macintyre PE, Huxtable CA, Flint SL, Dobbin MD. Costs and consequences: a review of discharge opioid prescribing for ongoing management of acute pain. Anaesth Intensive Care. 2014 Sep;42(5):558-74. doi: 10.1177/0310057X1404200504. PMID 25233168
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464
- [Background] Morris BJ, Mir HR. The opioid epidemic: impact on orthopaedic surgery. J Am Acad Orthop Surg. 2015 May;23(5):267-71. doi: 10.5435/JAAOS-D-14-00163. PMID 25911660
- [Background] Rodgers J, Cunningham K, Fitzgerald K, Finnerty E. Opioid consumption following outpatient upper extremity surgery. J Hand Surg Am. 2012 Apr;37(4):645-50. doi: 10.1016/j.jhsa.2012.01.035. Epub 2012 Mar 10. PMID 22410178
- [Background] Sabatino MJ, Kunkel ST, Ramkumar DB, Keeney BJ, Jevsevar DS. Excess Opioid Medication and Variation in Prescribing Patterns Following Common Orthopaedic Procedures. J Bone Joint Surg Am. 2018 Feb 7;100(3):180-188. doi: 10.2106/JBJS.17.00672. PMID 29406338
- [Background] Soffin EM, Waldman SA, Stack RJ, Liguori GA. An Evidence-Based Approach to the Prescription Opioid Epidemic in Orthopedic Surgery. Anesth Analg. 2017 Nov;125(5):1704-1713. doi: 10.1213/ANE.0000000000002433. PMID 29049115
- [Background] Tetrault JM, Butner JL. Non-Medical Prescription Opioid Use and Prescription Opioid Use Disorder: A Review. Yale J Biol Med. 2015 Sep 3;88(3):227-33. eCollection 2015 Sep. PMID 26339205